CLINICAL TRIAL: NCT05610982
Title: A Yoga Program for Adults Diagnosed With Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Brunet, Full Professor, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220544-01H
Record Dates: First submitted 2022-10-28; First posted 2022-11-09 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Survivorship; Cancer
Keywords: Yoga; Oncology; Hybrid/Bi-modal; Gynecologic Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga Program (Experimental): Participants will receive a yoga program program in-person or via real-time videoconferencing (if they choose).
  Interventions: Behavioral: Yoga Program

INTERVENTIONS:
Behavioral: Yoga Program — The yoga program involves two weekly 60-minute group-based classes. Participants can attend in-person or online (via Zoom). In total, 24 classes will be offered across 12 weeks. The program structure has been developed and approved by certified yoga instructors (n=12) and adults diagnosed with gynecologic cancer (n=6). The classes will follow a flexible base class that the instructor can then adapt as they see fit to promote participants' comfort, safety, and engagement. The program will also include group discussions and journaling that participants may participate in, if they choose. Finally, participants will be encouraged to access an online database of pre-recorded short-duration yoga practices to support their at-home practice.

SUMMARY:
Worldwide, >1.3 million adults are diagnosed with a gynecologic cancer each year. With rising survival rates, there are an increasing number of adults experiencing negative body image and decreased sexual functioning, resulting in reduced emotional, psychological, and social wellbeing and quality of life (QoL). It is vital that adults have access to programs focused on improving their body image and sexual functioning after a gynecologic cancer diagnosis. The Ottawa Regional Cancer Foundation (ORCF) is a non-for-profit, community-based organization offering support to persons with cancer. Strong university-community partnerships are essential to enhance translational and implementation research efforts. Stakeholders from academia, the healthcare sector, and the community (ORCF) are partnering to establish and implement an evidenced-based yoga program co-created with adults diagnosed with gynecologic cancer and yoga instructors to address the wellbeing needs of adults diagnosed with gynecologic cancer. The specific objectives of this mixed-methods feasibility trial are to: (1) evaluate the feasibility (recruitment, retention, adherence, intervention fidelity) of (a) the yoga program and (b) the trial methods the investigators propose to use to evaluate its benefits in a future trial (i.e., trial methods), (2) evaluate the acceptability of the yoga program and evaluative methods, and (3) explore preliminary effects of the program on key self-reported outcomes. Data will be used to frame evaluation and implementation efforts.

DETAILED DESCRIPTION:
Background: Each year, approximately 11, 000 women will be diagnosed with a gynecologic cancer in Canada (i.e., ovarian, endometrial/uterine, cervical, vulvar, vaginal). Despite rising survival rates, gynecologic cancer survivors report increased negative body image and decreased sexual functioning resulting in decreased quality of life. It is necessary to offer programs to help improve gynecologic cancer survivors' body image and sexual functioning, and thus enhance their quality of life. Previous research suggests that yoga can have a positive impact on body image and sexual functioning. Yoga, often referred to as a form of moving meditation, can help individuals shift their focus inward towards self-reflection, body appreciation, and gratitude whilst shifting their focus away from daily stressors. Moreover, yoga has the potential to be inclusive for those experiencing diminished physical capacities, such as cancer survivors, because there are many variations and modifications available for common poses. Further, yoga can be practiced in studio or at home with little to no equipment. Traditionally, yoga programs are developed based on researcher opinion and available resources (e.g., time, financial), resulting in a large variability in the length, duration, dosage, location, poses, and delivery-style of yoga sessions. This is problematic because it provides little insight into the type of yoga program that can optimize positive psychosocial outcomes (e.g., body image, sexual functioning) and the program components deemed beneficial to gynecologic cancer survivors. Further, instructors may (in)advertently contribute positively or negatively via authentic leadership, verbal commentary about weight and shape, social support, a culture of inclusion, and teasing. Despite the potential benefits of yoga, there are numerous pitfalls that may cause a yoga program to fail. Therefore, the specific objectives of this mixed-methods feasibility trial are to: (1) evaluate the feasibility (recruitment, retention, adherence, intervention fidelity) of (a) the yoga program and (b) the trial methods the investigators propose to use to evaluate its benefits in a future trial (i.e., trial methods), (2) evaluate the acceptability of the yoga program and evaluative methods, and (3) explore preliminary effects of the program on key self-reported outcomes. Data will be used to frame evaluation and implementation efforts.

Methods: Adults diagnosed with gynecologic cancer will be recruited from the Ottawa area. After obtaining informed consent verbally, participants will be randomized to a -3, -4 or -5 week baseline (control) A phase, and on a weekly basis for 3, 4, or 5 weeks (depending on group allocation), they will receive an email (at around the approximate same day/time to maintain equal spacing in-between assessments) with a link to a secure site to complete their online weekly assessment. For the intervention B phase, participants will take part in the 12-week yoga program and will be asked to complete assessments after the first class, after the 12th class (i.e., mid-point of program), and after completing their final class. For the follow-up A phase, participants will be asked to complete assessments 1, 4, and 8 weeks after their last class. They will be asked to complete all assessments within 48 hours of receiving the link; as it will expire after 48 hours, they will receive one email reminder 24 hours prior to expiration. Participants will also be invited to take part in an acceptability interview in-person (at the University of Ottawa or the ORCF) or via Microsoft Teams 1 week after their last class.

Discussion: Feasibility and acceptability data will help determine if/what changes/modifications are needed to improve the trial protocol and/or program, and will inform the timeline for a definitive trial. The psychosocial data collected will inform sample size calculation for a future RCT that aims to test the effects of this program in adults diagnosed with gynecologic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Have received a diagnosis of non-metastatic gynecologic cancer,
* Are able to read/speak/understand English,
* Have access to the Internet and an audio-visual device (e.g., computer, smart phone),
* Able and willing to travel to the Ottawa Regional Cancer Foundation twice a week for the first 2 weeks of the program.

Exclusion Criteria:

* Be non-ambulatory (i.e., unable to walk or require the assistance of a mobility device),
* Currently practicing yoga at least 1/week or have practiced consistently in the last 6 months (i.e., 1/week for 8 weeks).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-06-18 (Actual)

PRIMARY OUTCOMES:
Recruitment rates | Duration of study (12 months)
  The number of individuals who consent to participate in the study out of those who are assessed for eligibility
Study retention rates | Duration of study (12 months)
  How many participants complete follow-up assessments, with the primary endpoint at the final assessment at week 20
Program adherence rates | Duration of study (12 months)
  How many group-based classes participants attended, either in-person or online
Instructor fidelity to the program | Duration of study (12 months)
  The yoga classes will be recorded. At the cessation of the program, the recorded classes will be compared to the protocol for the classes (i.e., the sequence of poses and timing) to see how well the instructor adhered to the pre-determined protocol.
Participant engagement with group discussions | Duration of study (12 months)
  How often participants attended and interacted with other participants during group discussions.
Participant engagement with journaling | Duration of study (12 months)
  How many journal entries participants completed.
Participant engagement with pre-recorded practices | Duration of study (12 months)
  How many pre-recorded practices did participants watch and how often.
Acceptability of trial and program - Participants | At week 12
  Participants will be invited to complete semi-structured interviews to share their experiences, thoughts, and perspectives on (1) relevance of the program overall and its specific features, (2) suitability of the program overall and its specific features, (3) perceived benefits of the program overall and its specific features, (4) problems/concerns experienced during the program, and (5) suitability and problems/concerns with trial methods.
Acceptability of trial and program - Instructor | At week 12
  The yoga instructor will be asked to complete a semi-structured interview to explore their experiences delivering the intervention, as well as their thoughts about the content of the program, training and ongoing supervision, using the program manual, conducting classes, maintaining fidelity to the manual, and their motivation and confidence to conduct the program.

SECONDARY OUTCOMES:
Quality of life | Baseline (weekly for 3-5 weeks), program (week 1, week 6, week 12), and follow-up (week 13, week 16, week 20)
  Functional assessment of cancer therapy - General is a 27-item questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. The scale range is 0 (lowest) to 4 (highest) with a higher score meaning a higher quality of life.
Cognitive functioning | Baseline (weekly for 3-5 weeks), program (week 1, week 6, week 12), and follow-up (week 13, week 16, week 20)
  Perceived Cognitive Abilities sub-scale of the Functional Assessment of Cancer Therapy - Cognitive Function. The scale range is 0 (lowest) to 4 (highest) with a score meaning a higher perceived cognitive abilities.
Fatigue | Baseline (weekly for 3-5 weeks), program (week 1, week 6, week 12), and follow-up (week 13, week 16, week 20)
  Functional Assessment of Chronic Illness Therapy - Fatigue Scale. The scale range is 0 (lowest) to 4 (highest) with a higher score meaning a higher level of fatigue.
Feelings and problems regarding sexuality | Baseline (weekly for 3-5 weeks), program (week 1, week 6, week 12), and follow-up (week 13, week 16, week 20)
  Female Sexual Distress Scale-Revised. The scale range is 0 (lowest) to 4 (highest) with a higher score meaning a higher level of sexual distress.
Body image | Baseline (weekly for 3-5 weeks), program (week 1, week 6, week 12), and follow-up (week 13, week 16, week 20)
  Body Image Scale. The scale range is 1 (lowest) to 4 (highest) with a higher score meaning a higher level of negative body image.
Perceived stress | Baseline (weekly for 3-5 weeks), program (week 1, week 6, week 12), and follow-up (week 13, week 16, week 20)
  Perceived Stress Scale. The scale range is 0 (lowest) to 4 (highest) with a higher score meaning a higher level of perceived stress.
Psychological flexibility | Baseline (weekly for 3-5 weeks), program (week 1, week 6, week 12), and follow-up (week 13, week 16, week 20)
  Acceptance and Action Questionnaire II. The scale range is 1 (lowest) to 7 (highest) with a higher score meaning a higher level of psychological inflexibility.
Embodiment | Baseline (weekly for 3-5 weeks), program (week 1, week 6, week 12), and follow-up (week 13, week 16, week 20)
  Experiences of Embodiment Scale. The scale range is 1 (lowest) to 5 (highest) with a higher score meaning a higher level of embodiment.

OTHER OUTCOMES:
Sociodemographic and medical characteristics | Baseline (week 0)
  Self-reported socio-demographic and medical information (e.g., age, gender, civil and educational status, ethnicity) will be collected and used to describe the sample. Participants will be provided with a range of response options for each item

CONTACTS AND LOCATIONS:
Overall Officials: Jenson Price, PhD c, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Wagner, L.I., et al., Measuring patient self-reported cognitive function: development of the functional assessment of cancer therapy-cognitive function instrument. J Support Oncol, 2009. 7(6): p. W32-W39.
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Derogatis L, Clayton A, Lewis-D'Agostino D, Wunderlich G, Fu Y. Validation of the female sexual distress scale-revised for assessing distress in women with hypoactive sexual desire disorder. J Sex Med. 2008 Feb;5(2):357-64. doi: 10.1111/j.1743-6109.2007.00672.x. Epub 2007 Nov 27. PMID 18042215
- [Background] Hopwood P, Fletcher I, Lee A, Al Ghazal S. A body image scale for use with cancer patients. Eur J Cancer. 2001 Jan;37(2):189-97. doi: 10.1016/s0959-8049(00)00353-1. PMID 11166145
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Hardin EE, Lakin JL. The Integrated Self-Discrepancy Index: a reliable and valid measure of self-discrepancies. J Pers Assess. 2009 May;91(3):245-53. doi: 10.1080/00223890902794291. PMID 19365765
- [Background] Piran N, Teall TL, Counsell A. The experience of embodiment scale: Development and psychometric evaluation. Body Image. 2020 Sep;34:117-134. doi: 10.1016/j.bodyim.2020.05.007. Epub 2020 Jun 14. PMID 32554242
- [Derived] Price J, Sabir S, Westlake B, Brunet J. The impact of a co-created yoga program for women diagnosed with gynecologic cancer on patient-reported outcomes: a series N-of-1 trial. Support Care Cancer. 2026 Jan 10;34(2):80. doi: 10.1007/s00520-025-10279-1. PMID 41518418
- [Derived] Price J, Brunet J. A single-subject research design evaluating a co-created yoga program for adults with gynecologic cancer: feasibility study protocol. Pilot Feasibility Stud. 2024 Jan 16;10(1):8. doi: 10.1186/s40814-023-01435-7. PMID 38229143